



Bath BA2 7AY · United Kingdom

Telephone +44 (0)1225 383843 Facsimile +44 (0)1225 386752 Email psychology-enquiries@bath.ac.uk

9

www.bath.ac.uk/psychology

Chief Investigator: Emil Vuillermoz

ev329@bath.ac.uk

IRAS ID: 318755

## **FULL STUDY TITLE:**

Acceptability and preliminary effectiveness of a mobile health intervention (Untire app) for adult cancer patients and survivors with cancer related fatigue: A pilot clinical study

## **SHORT TRIAL TITLE:**

Acceptability of an updated version of the Untire mHealth app.

RESEARCH REFERENCE NUMBERS

**IRAS Number: 318755** 

Clinical trials.gov Number: [not yet assigned]

REC reference: 23/YH/0101

Date created: 22/10/2022 Date reviewed:05/05/2023





Bath BA2 7AY · United Kingdom

Telephone +44 (0)1225 383843 Facsimile +44 (0)1225 386752 psychology-enquiries@bath.ac.uk

www.bath.ac.uk/psychology

IRAS ID: 318755

Chief Investigator: Emil Vuillermoz

ev329@bath.ac.uk

## **Informed Consent**

Study title: Acceptability and preliminary effectiveness of a mobile health intervention (Untire app) for adult cancer patients and survivors with cancer related fatigue: A pilot clinical study

Chief Investigator: **Emil Vuillermoz** Research Supervisor: Dr Cara Davis

> if you agree, please type your initials into each box

| | initial | s into each box |
|---|---|---|
| 1. | I confirm that I have read the participant information page dated 29/04/23 (version 1.3) for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I am aware that participation is voluntary. I understand that I can decide at any time not to participate after all or to withdraw from the study. Withdrawing from this study will not negatively impact the quality of care I receive from the NHS. | |
| 3. | I agree for a member of the research team to contact me (using the contact details I provided) to ask about my experience of using the Untire app. This would include if I chose to stop using the app at any point. | |
| 4. | I understand that this study will require access to my data. This includes data from questionnaires I fill in, data that I enter into the app and stored automatically regarding my app use. This will only be accessed by the research team. | |
| 5. | I agree that my data will remain confidential and only be accessed by members of the research team. My data will be stored at the University of Bath for 5 years after the study. | |
| 6. | I agree to the use of anonymised quotes I might give to be used in research reports and publications. | |
| 7. | I agree to take part in this study. | |

Date created: 22/10/2022 Date reviewed:05/05/2023







Bath BA2 7AY · United Kingdom

Telephone +44 (0)1225 383843 Facsimile +44 (0)1225 386752 Email

psychology-enquiries@bath.ac.uk www.bath.ac.uk/psychology

IRAS ID: 318755

Chief Investigator: Emil Vuillermoz ev329@bath.ac.uk

| Additio | onal | | |
|---|---|---|---|
| 8. | 3. [Optional] I agree to be contacted in the future about ethically approved research studies for which I may be suitable. I understand that agreeing to be contacted does not oblige me to participate in any further studies. | | |
| | Name: Contact number /email: | | |
| I hereby | y declare that I have | been fully informed ab | out this study. |
| Name o | of Participant | Date | Signature |
| Name o | of Person taking | Date | Signature |

A copy of this signed consent form will be kept by the chief investigator and stored digitally on a secure research data storage drive (X:Drive) at the University of Bath. This consent form will be stored separately from any study data (Questionnaires). It is advised that you also retain a copy of your signed consent form.

Date created: 22/10/2022 Date reviewed:05/05/2023